CLINICAL TRIAL: NCT01741142
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of ABT-436 in Major Depressive Disorder
Brief Title: Efficacy and Safety Study of ABT-436 in Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision based on strategic determination; not safety.
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-733
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-436 (Experimental): Subject receiving ABT-436
  Interventions: Drug: ABT-436
- Escitalopram (Active Comparator): Subject receiving escitalopram.
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Subject receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-436 — Subjects receiving ABT-436
  Arms: ABT-436
Drug: Escitalopram — Subjects receiving escitalopram
  Arms: Escitalopram
Drug: Placebo — Subject receiving placebo
  Arms: Placebo

SUMMARY:
The purpose is to study the efficacy and safety of ABT-436 in Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision diagnosis of major depressive disorder without psychotic features
* No current antidepressant treatment within 7 half-lives or 2 weeks, whichever is longer, prior to Day minus 1.
* Can safely be treated on an outpatient basis.
* A condition of general good physical health.
* Surgically sterile, using a highly effective method of birth control or (if female) at least 1 year post menopausal.

Exclusion Criteria:

* History of hypersensitivity, intolerance or adverse reaction to escitalopram that led to discontinuation, or hypersensitivity to citalopram. History of serotonin syndrome.
* Inadequate response to more than two different antidepressant medications during the current major depressive episode.
* History of electroconvulsive therapy, vagal nerve stimulation or deep brain stimulation.
* History of transcranial magnetic stimulation during the current major depressive episode.
* Psychotherapy that has not been ongoing for at least 3 months prior to Day minus 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy variable will be change from baseline to Week 6 visit on Montgomery-Asberg Depression Rating Scale (MADRS) total score. | Week 6
  Primary efficacy variable will be change from baseline to Week 6 visit on Montgomery-Asberg Depression Rating Scale (MADRS) total score.

SECONDARY OUTCOMES:
Secondary efficacy variables include change from Baseline to Week 6 on clinician-rated Hamilton Depression Rating Scale. | Week 6
  Secondary efficacy variables include change from Baseline to Week 6 on clinician-rated Hamilton Depression Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Rendenbach-Mueller, PhD, Study Director — AbbVie
Locations (18):
- United States (18):
  - Site Reference ID/Investigator# 85593, Little Rock, Arkansas
  - Site Reference ID/Investigator# 87228, Garden Grove, California
  - Site Reference ID/Investigator# 87214, National City, California
  - Site Reference ID/Investigator# 87220, Oakland, California
  - Site Reference ID/Investigator# 87215, Bradenton, Florida
  - Site Reference ID/Investigator# 87225, South Miami, Florida
  - Site Reference ID/Investigator# 85594, Atlanta, Georgia
  - Site Reference ID/Investigator# 85580, Marlton, New Jersey
  - Site Reference ID/Investigator# 87227, Brooklyn, New York
  - Site Reference ID/Investigator# 87223, New York, New York
  - Site Reference ID/Investigator# 87217, Dayton, Ohio
  - Site Reference ID/Investigator# 87226, Portland, Oregon
  - Site Reference ID/Investigator# 87221, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 87219, Austin, Texas
  - Site Reference ID/Investigator# 87216, Dallas, Texas
  - Site Reference ID/Investigator# 87933, Houston, Texas
  - Site Reference ID/Investigator# 88874, Salt Lake City, Utah
  - Site Reference ID/Investigator# 88876, Seattle, Washington